CLINICAL TRIAL: NCT05557448
Title: An Exploratory Study to Evaluate the Efficacy and Safety of TYNADOTE® Combined N-acetylcysteine in the Treatment of Acetaminophen Overdose
Brief Title: To Evaluate the Efficacy and Safety of TYNADOTE® in the Treatment of Acetaminophen Overdose
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sinew Pharma Inc. (Industry)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TYNADOTE-2-001
Record Dates: First submitted 2022-09-22; First posted 2022-09-28 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Hepatitis
Keywords: Paracetamol; Acetaminophen; Acute liver failure; N-acetylcysteine; Acetaminophen overdose
MeSH Terms: conditions — Hepatitis; Liver Failure, Acute

STUDY DESIGN:
Intervention Model Description: test drug
Who Masked: Participant, Investigator
Masking Description: placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test drug (Active Comparator): 200 mg/every 4 hours, with a loading dose (400 mg) and then followed by 17 maintenance doses
  Interventions: Drug: TYNADOTE
- Placebo (Placebo Comparator): 200 mg/every 4 hours, with a loading dose (400 mg) and then followed by 17 maintenance doses
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: TYNADOTE — Subjects will take 200 mg/every 4 hours, with a loading dose (400 mg) and then followed by 17 maintenance doses
  Arms: Test drug
Drug: Placebo Oral Tablet — Subjects will take 200 mg/every 4 hours, with a loading dose (400 mg) and then followed by 17 maintenance doses
  Arms: Placebo

SUMMARY:
To evaluate the efficacy and safety of TYNADOTE® in the treatment of acetaminophen overdose

DETAILED DESCRIPTION:
This will be a 21-day study to evaluate the efficacy and safety of TYNADOTE® in the treatment of acetaminophen overdose.

After the inform consent is obtained from the subject or his/her legal guardians, the designated assessment will be performed. Subjects who fulfill all the inclusion and exclusion criteria will be eligible to enter the study. Except standard NAC antidote therapy, subjects would be randomized as 1:1 ratio to combine oral TYNADOTE® or placebo.

Eligible subjects will be randomized to receive oral TYNADOTE®/placebo combined iv NAC, and the regimen was listed as below:

The NAC intravenous loading dose is 150 mg/kg over a period of 15 to 60 minutes, followed by an infusion of 12.5 mg/kg per hour over a 4-hour period, and finally an infusion of 6.25 mg/kg per hour over a 16-hour period. Study drug, TYNADOTE® /placebo, should be given a loading dose of 400 mg, followed by 17 maintenance doses of 200 mg every 4 hours (Day 1 to Day 3).

During the treatment period, vital signs will be checked 15 minutes prior to dosing, 30 minutes, 60 minutes, then 2, 4, 8, 12, 24, 36, 48, 60 and 72 hours after first dosing. Blood samples will be collected for liver injuries and function test, including AST, ALT, total bilirubin, direct bilirubin and prothrombin time (INR), prior to dosing, 4 hours, 12 hours, 24 hours, 36 hours, 48 hours, 60 hours, 72 hours after first dosing. Blood samples for drug/metabolites concentration, including TYNADOTE® plasma concentration (trough level), plasma acetaminophen concentration, AAP-Cys and AAP-Cys adducts concentration, prior to dosing, 4 hours, 12 hours, 24 hours, 36 hours, 48 hours, 60 hours and 72 hours after first dosing. Blood samples for biochemistry and hematology, Day 1-3.

After completing the treatment (Day 3), subject will conduct the following evaluations before discharge:

* Review of adverse events
* Review of concomitant medications
* Physical examination On Day 7 and Day 21, subjects should return to the clinics for liver injuries/function follow up and reviewing the adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Poisoning and hospitalized patients taking acetaminophen.
* Acute ingestion of more than 150 mg/kg or plasma concentration of Acetaminophen is above the treatment line on single acute acetaminophen overdose nomogram.
* Male or female with age more than 20 years at Screening.
* Ability and willingness to provide informed consent, adhere to the study visit schedule and complete all study assessments.

Exclusion Criteria:

* Subjects with Sequential Organ Failure Assessment (SOFA) Score higher than 12.
* Subjects who fulfilled the King's College Hospital (KCH) Criteria for liver transplantation.
* Subjects who was conscious disturbance.
* History of allergic response(s) to N-acetylcysteine (NAC), mannitol, sucralose or related drugs.
* Subject who was unable to take medicine by oral route.
* Receiving any investigational drug within 30 days prior to first dosing.
* Subject who had attacked asthma or bronchitis combined with medication therapy within six months prior to enrollment.
* Donating greater than 150 mL of blood within two months prior to first dosing or donating plasma (e.g. plasmapheresis) within 14 days prior to first dosing. All subjects will be advised not to donate blood for four weeks after completing the study.
* Subject is pregnant or breastfeeding. Women of childbearing potential must have a negative serum pregnancy test at baseline.
* Anuria, pulmonary congestion, severe congestive heart failure, brain hemorrhage, or any conditions that in the opinion of the investigator may interfere with the evaluation of study objectives.
* The combination of poisoning contains acetaminophen and other compound.
* Body weight less than 50 kg.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Alanine aminotransferase | Day 3
  Percentage change from baseline of ALT at Day 3.

SECONDARY OUTCOMES:
Alanine aminotransferase | Day 7
  Percentage change from baseline of ALT at Day 7
Alanine aminotransferase | Day 7
  Percentage change from baseline of AST at Day 3, Day 7
Total bilirubin | Day 3, Day 7 and Day 21
  Incidence of total bilirubin > 2.5mg/dL at Day 3, Day 7, Day 21
Inte- rnational Normalize Ratio | Day 3, Day 7 and Day 21
  Incidence of INR > 1.25 at Day 3, Day 7, Day 21
Aspartate aminotransferase or Alanine aminotransferase | Day 3, Day 7 and Day 21
  Incidence of AST or ALT >1000 U/L at Day 3, Day 7, Day 21
Hepatic failure rate (hepatic encephalopathy, ascites, total bilirubin, INR or liver transplantation) | Day 7 and Day 21
  Hepatic failure rate (hepatic encephalopathy, ascites, total bilirubin >2.5mg/dL, INR >1.25, or liver transplantation) at Day 7, Day 21
Mortality rate | Day 7 and Day 21
  Mortality rate at Day 7, Day 21
Free plasma acetaminophen-cysteine (AAP-Cys) and AAP-Cys adducts | Day 1-3
  The time-interval weighted area under the curve (AUC) of free plasma acetaminophen-cysteine (AAP-Cys) and AAP-Cys adducts within 72-hour treatment period
TYNADOTE® plasma concentration | Day 1-3
  The time-interval weighted area under the curve (AUC) of TYNADOTE® plasma concentration during 72-hour treatment period

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Beitou District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided